CLINICAL TRIAL: NCT02065388
Title: Pharmacogenetic Dosing of Warfarin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Academia Sinica, Taiwan (Other)
Collaborators: Chang Gung Memorial Hospital (Other); China Medical University Hospital (Other); Kaohsiung Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AS-IRB01-100070
Record Dates: First submitted 2014-02-09; First posted 2014-02-19 (Estimated); Last update posted 2014-02-19 (Estimated); Status verified 2014-02

CONDITIONS: Stroke; Venous Thrombosis; Atrial Fibrillation; Atrial Flutter
MeSH Terms: conditions — Stroke; Venous Thrombosis; Atrial Fibrillation; Atrial Flutter | interventions — Warfarin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Standard of care dosing for warfarin (Active Comparator): Loading dose (5mg) of warfarin for the first 3 days of treatment. Dose adjustment after initiation will using guideline modified from Tait el al. (1998).
  Interventions: Behavioral: Standard of care dosing for warfarin
- Genotype-guided dosingTaiwan algorithm for warfarin (Experimental): Initial loading dosing of warfarin for the first 3 days of treatment will be determined by the Taiwan algorithm that uses clinical and genetic information. Dose adjustment after initiation will using guideline modified from Tait el al. (1998).
  Interventions: Genetic: Genotype-guided dosingTaiwan algorithm for warfarin
- Genotype-guided dosing IWPC algorithm for warfarin (Experimental): Initial loading dosing of warfarin for the first 3 days of treatment will be determined by the IWPC algorithm that uses clinical and genetic information. Dose adjustment after initiation will using guideline modified from Tait el al. (1998).
  Interventions: Genetic: Genotype-guided dosing IWPC algorithm for warfarin

INTERVENTIONS:
Behavioral: Standard of care dosing for warfarin
  Arms: Standard of care dosing for warfarin
Genetic: Genotype-guided dosingTaiwan algorithm for warfarin
  Arms: Genotype-guided dosingTaiwan algorithm for warfarin
Genetic: Genotype-guided dosing IWPC algorithm for warfarin
  Arms: Genotype-guided dosing IWPC algorithm for warfarin

SUMMARY:
Purpose:

Warfarin is now the most commonly used oral anticoagulant. This drug has inter-individual variability due to the genetic polymorphisms in the warfarin metabolizing enzyme, CYP2C9 and warfarin target, VKORC1. The investigators' team developed a pharmacogenetic dosing algorithm which can predict patients required warfarin dose, thus could prevent warfarin induced warfarin adverse events.

Methods:

The investigators recruited patients with indications for warfarin, the genotypes of VKORC1 and CYP2C9 were determined by the hospitals and verified by National Center for Genome Medicine. The investigators then randomized the patients to one of three arms: 1. Warfarin dose predicted by dosing algorithm developed by the International Warfarin pharmacogenetic Consortium (IWPC), 2. Algorithm developed by the Taiwan Warfarin Consortium and 3. Standard of care. The investigators aimed to determine whether using genetic dosing algorithm can lead to more stable dose and safer use of the drug.

ELIGIBILITY:
Inclusion Criteria:

* Patients must give their informed consent and complete the case report form.
* Patients must be over the age of 20.
* Patients have clinical indications for warfarin therapy but do not have any prior warfarin treatment.

Exclusion Criteria:

* Patients who did not complete the informed consent form or the CRF
* Patients who are less than the age of 20.
* Patients who had prior or is currently on warfarin treatment.
* Patients who have hemorrhagic tendencies or hemorrhagic diseases defined as copious bleeding caused by viral or bacterial infections; cancer and hepatic dysfunction defined as GOP and GPT values three times higher than normal value
* Patients who has Vitamin K deficiency
* Female patients who is currently pregnant

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2009-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Time spent in target INR range | first month of therapy
  time spent in target INR range Time in the target INR Range will be the primary endpoints because of its strong association with adverse events: patients with subtherapeutic INR values are at increased risk of thrombosis and patients with high INR values are at increased risk of hemorrhage during warfarin treatment initiation.

CONTACTS AND LOCATIONS:
Overall Officials: Ming Ta Michael Lee, PhD, Principal Investigator — Institute of Biomedical Sciences, Academia Sinica
Locations (3):
- Taiwan (3):
  - Kaohsiung Medical University, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Chang Gung Memorial Hospital, Taoyuan District

REFERENCES:
- [Derived] Ohara M, Takahashi H, Lee MT, Wen MS, Lee TH, Chuang HP, Luo CH, Arima A, Onozuka A, Nagai R, Shiomi M, Mihara K, Morita T, Chen YT. Determinants of the over-anticoagulation response during warfarin initiation therapy in Asian patients based on population pharmacokinetic-pharmacodynamic analyses. PLoS One. 2014 Aug 22;9(8):e105891. doi: 10.1371/journal.pone.0105891. eCollection 2014. PMID 25148255